CLINICAL TRIAL: NCT01970917
Title: Effect of Olixia Pure® Eye Drops on Tear Film Thickness in Healthy Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. PD Dr., Medical University of Vienna
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Basic Science
Other Study IDs: OPHT-190313
Record Dates: First submitted 2013-07-11; First posted 2013-10-28 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Dry Eye Syndrome; Healthy
Keywords: tear film thickness; optical coherence tomography; topical lubricants; tear film thickness in healthy subjects
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Healthy volunteers right eye (Other): The medical device will be randomly assigned to the right or left eye on the study day (randomization 1:1) whereas the fellow eye will receive placebo.
  Interventions: Device: Olixia pure eye drops; Device: Placebo
- Healthy volunteers left eye (Other): The medical device will be randomly assigned to the right or left eye on the study day (randomization 1:1) whereas the fellow eye will receive placebo.
  Interventions: Device: Olixia pure eye drops; Device: Placebo

INTERVENTIONS:
Device: Olixia pure eye drops
Device: Placebo — 0.9% physiological saline solution

SUMMARY:
Dry eye syndrome (DES) is a common ocular disease, especially in the elderly population. Despite many treatment approaches, instillation of topical lubricants remains the mainstay of therapy. However, most of the topical lubricants available are not very well characterized and data about efficacy is sparse.

The aim of the present project is to investigate the effect of topically administered Olixia pure® eye drops on tear film thickness in healthy subjects.

Tear film thickness will be determined using ultra high-resolution optical coherence tomography (OCT). Measurements will be performed before instillation of the eye drops and every 10 minutes after instillation for one hour. One eye will receive Olixia pure® eye drops, the fellow eye will receive physiologic saline solution as placebo control. The study eye will be chosen randomly.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged over 18 years
* Normal findings in the medical history unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, ametropia < 6 Dpt.
* Schirmer I test > 10 mm and BUT > 10 sec

Exclusion Criteria:

* Regular use of medication (except contraceptives), abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Treatment in the previous 3 weeks with any drug
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Ametropia =/> 6 Dpt
* Pregnancy
* Difference of more than 5 mm in Schirmer I test or difference of > 3 sec in BUT between the two eyes
* Known medical history of allergy, hypersensitivity or poor tolerance to any components of the medication or medical product used in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Tear film thickness | up to one hour

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Garhoefer, MD, Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Vienna, Vienna, Austria